CLINICAL TRIAL: NCT05524090
Title: Nationwide Implementation Program for Optimal Multidisciplinary Management and Resection of Locally Advanced Pancreatic Cancer (PREOPANC-4)
Brief Title: PREOPANC-4 Implementation Program for Locally Advanced Pancreatic Cancer
Acronym: PREOPANC-4
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: UMC Utrecht (Other); Erasmus Medical Center (Other); Leiden University Medical Center (Other); University Medical Center Groningen (Other); Radboud University Medical Center (Other); Maastricht University Medical Center (Other); Medisch Spectrum Twente (Other); Isala (Other); Frisius Medisch Centrum (Other); Onze Lieve Vrouwe Gasthuis (Other); Amphia ziekenhuis (Unknown); Jeroen Bosch Ziekenhuis (Other); Catharina Ziekenhuis Eindhoven (Other); University of Colorado, Denver (Other); Heidelberg University (Other); M.D. Anderson Cancer Center (Other); NYU Langone Health (Other); Dutch Cancer Society (Other); Maag Lever Darm Stichting (Other); Deltaplan Alvleesklierkanker (Unknown)
Responsible Party: Principal Investigator, M.G. Besselink, prof. dr. M.G. Besselink, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W21_487 # 21.541
Record Dates: First submitted 2022-08-16; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Pancreatic Cancer; Locally Advanced Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma Non-resectable; Chemotherapy Effect
Keywords: Nationwide implementation International Best-Practice; The Netherlands; International Best-Practice; Patient Selection; Patient-centered
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Implementation cohort: Inclusion criteria:
  1. Age ≥18 years;
  2. Pathology confirmed LAPC*;
  3. CT-based non-progressive disease in accordance with the RECIST criteria after at least 4 months of systemic chemotherapy ([m]FOLFIRINOX or gemcitabine-nab-paclitaxel).
  Exclusion criteria:
  (1) Metastatic pancreatic cancer prior to induction chemotherapy.
  *According to the Dutch Pancreatic Cancer Group (DPCG) definition: >90 degrees arterial tumor involvement (i.e. superior mesenteric artery, celiac axis, and/or hepatic artery) and/or portovenous involvement of either >270 degrees or occlusion.
  Interventions: Other: Implementation - International best-practice care

INTERVENTIONS:
Other: Implementation - International best-practice care — The PREOPANC-4 project aims to safely implement the international standard of excellence for LAPC management and surgery using a multidisciplinary best-practice training program, based on the experiences of four leading international expert centers (i.e. NYU Langone Health, University of Colorado, Heidelberg University, and MD Anderson Cancer Center). We hypothesize that the PREOPANC-4 implementation project will result in the improvement in multidisciplinary patient management and selection in line with current international best-practice.

SUMMARY:
A prospective, nationwide, implementation program of the international standard of excellence for locally advanced pancreatic cancer (LAPC) care in the Netherlands (2021[7]-2030[6]), including a multidisciplinary training program by the four leading international expert centers.

The PREOPANC-4 project aims a safe and patient-centered implementation of the international standards of excellence for LAPC (surgery) in the Netherlands.

DETAILED DESCRIPTION:
Rationale:

Non-metastasized locally advanced pancreatic cancer (LAPC) is diagnosed in 35% of all pancreatic cancer patients and is traditionally treated with palliative care. Recently, the multidisciplinary management of LAPC has evolved by the introduction of modern multi-agent induction chemotherapies, leading to an increased resection rate and improved outlook for five-year survival. In contrast, five-year survival after chemotherapy without surgery is virtually non-existent. In the Netherlands, the LAPC resection rate after induction chemotherapy remains low with 8% versus 25% in international centers of excellence, leading to missed opportunities for five-year survival in a selected subgroup of LAPC patients. Explanations for this large difference include the spectrum of chemotherapy use, interpretation of diagnostics, patient selection, and surgical techniques.

Objective:

A safe and patient-centered implementation of the international standards of excellence for LAPC (surgery) in the Netherlands.

Study design:

A prospective, nationwide, implementation program of the international standard of excellence for LAPC care in the Netherlands (2021[7]-2030[6]), including a multidisciplinary training program by the four leading international expert centers (i.e. University of Heidelberg, University of Colorado, NYU Langone, and MD Anderson Cancer Center). Subsequently, the three Dutch centers with the highest surgical volume and documented experience in LAPC surgery will implement this highly complex LAPC surgery in close collaboration with the other Dutch Pancreatic Cancer Group (DPCG) centers. Patients who meet the inclusion criteria will be discussed within an online (inter)national expert panel to properly select patient for surgery. In addition, the other DPCG centers can present their LAPC patients to this panel for advice about (surgical) treatment options and if these patients should be referred to the three high-volume DPCG centers for surgery. Outcomes will be compared with a historical Dutch LAPC cohort, using propensity score matching.

Study population:

Adult patients with pathology confirmed non-metastasized LAPC and non-progressive disease after at least four months of (modified) FOLFIRINOX or gemcitabine-nab-paclitaxel induction chemotherapy and fit for major surgery.

Study aim:

The primary study aim is to double the LAPC resection rate in the Netherlands from 8% to 16% with adequate survival and morbidity targets.

Primary targets:

1. Survival: After resection, mOS of 25 months, 1-year survival >90%, and 5-year survival >20%. These outcomes will be compared to the Dutch cohort of patients (2015-2020) with RECIST non-progressive LAPC after induction chemotherapy who did not undergo surgical exploration;
2. In-hospital morbidity and mortality: in-hospital/30-day mortality ≤5% and in-hospital major morbidity of <50% after resection, which will be compared with a recent Dutch cohort (2015-2020) of resected patients with borderline resectable and locally advanced pancreatic cancer after induction/neoadjuvant therapy.

Secondary targets:

1. Non-inferior radical resection (R0) rate as compared to a recent Dutch cohort (2015-2020) of resected patients with borderline resectable and locally advanced pancreatic cancer after induction/neoadjuvant therapy;
2. Non-inferior quality of life, mental and physical health status, and potential side effects on the long-term follow-up, compared to a control cohort of Dutch LAPC patients;
3. Non-inferior patients' healthcare satisfaction, compared to the Dutch historical cohort of pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Pathology-confirmed (LAPC)*
* CT-based non-progressive disease (RECIST criteria) after at least 4 months of systemic chemotherapy ([m]FOLFIRINOX / gemcitabine-nab-paclitaxel).

Exclusion Criteria:

* Metastatic pancreatic cancer prior to induction chemotherapy.

  * According to the Dutch Pancreatic Cancer Group (DPCG) definition: >90 degrees arterial tumor involvement (i.e. superior mesenteric artery, celiac axis, and/or hepatic artery) and/or portovenous involvement of either >270 degrees or occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with pathology confirmed non-metastasized LAPC and non-progressive disease after at least two months of (modified) FOLFIRINOX or gemcitabine-nab-paclitaxel induction chemotherapy and fit for major surgery.
Sampling Method: Probability Sample
Enrollment: 223 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Resection rate | Immediately after completing the inclusion period (December 31, 2024).
  Resection rate of the pancreatic tumor
Overall survival (OS) | After completing the follow-up period (December 31, 2029)
  OS from time of resection (mOS, 1-year OS & 5-year OS)
In-hospital mortality | Yearly assessment throughout the inclusion period
  Mortality after resection (during primary hospitalization)
In-hospital major morbidity | Yearly assessment throughout the inclusion period
  Clavien-Dindo grade IIIa or higher major morbidity after resection (during primary hospitalization)

SECONDARY OUTCOMES:
R0 resection rate | Immediately after completing the inclusion period (December 31, 2024).
  R0 (microscopic radical resection >1mm) versus R1 (microscopic residual tumor ≤1mm). NB. For the anterior margin, only direct ingrowth is considered as R1.
Quality of life | Measured at 3, 6, 9, 12, 18, and 24 months from diagnosis, followed by yearly measurements.
  EORTC QLQ-C30: global health status
  Outcome measures will be calculated, according to the validated questionnaire manuals.
Shared decision-making: patients' healthcare satisfaction | Measured at 3, 6, 9, 12, 18, and 24 months from diagnosis, followed by yearly measurements.
  APECC decision-making self-efficacy scale.
  Outcome measures will be calculated, according to the validated questionnaire manuals.

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Besselink, MD, MSc, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, locatie AMC, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Stoop TF, Seelen LWF, van 't Land FR, van der Hout AC, Scheepens JCM, Ali M, Stiggelbout AM, van der Kolk BM, Bonsing BA, Lips DJ, de Groot DJA, van Veldhuisen E, Kerver ED, Manusama ER, Daams F, Kazemier G, Cirkel GA, van Tienhoven G, Patijn GA, Lelieveld-Rier HN, de Hingh IH, van Hellemond IEG, Wijsman JH, Erdmann JI, Mieog JSD, de Vos-Geelen J, de Groot JWB, Lutchman KRD, Mekenkamp LJ, Kranenburg LW, Beuk LPM, Nijkamp MW, den Dulk M, Polee MB, Homs MYV, Wumkes ML, Stommel MWJ, Busch OR, de Wilde RF, Theijse RT, Luelmo SAC, Festen S, Bollen TL, Neumann UP, de Meijer VE, Draaisma WA, Groot Koerkamp B, Molenaar IQ, Wolfgang CL, Del Chiaro M, Katz MGH, Hackert T, Rietjens JAC, Wilmink JW, van Santvoort HC, van Eijck CHJ, Besselink MG; Dutch Pancreatic Cancer Group. Nationwide implementation of the international multidisciplinary best-practice for locally advanced pancreatic cancer (PREOPANC-4): study protocol. BMC Cancer. 2025 Feb 19;25(1):299. doi: 10.1186/s12885-025-13554-w. PMID 39972248